CLINICAL TRIAL: NCT03370146
Title: Can Mental Training Based on Motor Imagery Speed up the Rehabilitation of Walking? Efficacy of a Controlled Procedure and Neurofunctional Bases of Recovery in Patients With Total Knee Arthroplasty
Brief Title: Motor Imagery and Rehabilitation of Orthopaedic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: L3020
Record Dates: First submitted 2017-11-29; First posted 2017-12-12 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Cognitive Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TKA patients - Experimental Group
  Interventions: Behavioral: Mental training based on Motor Imagery; Behavioral: Evaluation of gait abilities
- TKA patients - Control Group 1
  Interventions: Behavioral: Cognitive training; Behavioral: Evaluation of gait abilities
- Healthy subjects - Control Group 2
  Interventions: Behavioral: Evaluation of gait abilities

INTERVENTIONS:
Behavioral: Mental training based on Motor Imagery — Patients of the experimental group will be instructed to imagine walking, from a first person perspective, focusing on the kinaesthetic sensations typically associated with the movement. The motor imagery training will be performed using the support of a laptop, on which there will be presented complex static scenes, representing different kind of paths with different landmarks to reach during the mental walking.
  Groups: TKA patients - Experimental Group
Behavioral: Cognitive training — Patients of the control group 1 will undergo a general cognitive training, not based on motor imagery.
  Groups: TKA patients - Control Group 1
Behavioral: Evaluation of gait abilities — All the subjects included in the trial will undergo a series of behavioral test for the evaluation of gai abilities

SUMMARY:
Motor imagery is increasingly used as a plasticity-booster to complement conventional rehabilitation. Here the investigators test the hypothesis that the combination of mental training with conventional rehabilitation may speed up the recovery in patients with total knee arthroplasty. The investigators also characterize the brain correlates of such recovery with imagery tasks for virtual reality environments.

ELIGIBILITY:
Inclusion Criteria:

* Right handed
* No contraindication to the fMRI exam

Exclusion Criteria:

* Contraindication to the fMRI exam

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experimental group (MI training): 24 candidates to TKA (aged between 45 and 65 years) will undergo a specific MI training during the period of post-surgical rehabilitation, in addition to the usual physical rehabilitation.
  Control group 1 (non-specific cognitive training): 24 candidates to TKA will undergo a non-specific cognitive treatment during the period of post-surgical rehabilitation, in addition to the usual physical rehabilitation.
  Control group 2: 48 subjects with similar demographic characteristics to those of the previous two groups will be evaluated with the same cognitive/fMRI paradigm to assess in TKA candidates the presence of anomalies of cortical organization of the motor system in the pre-surgical phase.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03-17 (Actual); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Speed of walking | 20 days
  The speed of walking recorded in total knee arthroplasty patients of the experimental group will be compared with the same measure recorded in both control groups.
BOLD (blood oxygen level-dependent) activity | 20 days
  The BOLD activity recorded during functional magnetic resonance imaging (fMRI) in TKA patients of the experimental group will be compared with the same measure recorded in both control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Galeazzi Orthopedic Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No